CLINICAL TRIAL: NCT06826222
Title: The Effect of Sodium Bicarbonate Intake on Endurance Performance in Recreational Female Runners
Brief Title: Sodium Bicarbonate Intake on Endurance Performance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Selin Aktitiz, Research Assistant, Hacettepe University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: KA-24026
Record Dates: First submitted 2025-02-10; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: The Effects of Sodium Bicarbonate Supplementation on Endurance Performance in Recreational Female Runners
Keywords: Sodium Bicarbonate; Female Athletes; Endurance Performance; Running; Buffering Capasity
MeSH Terms: interventions — Sodium Bicarbonate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double Blind Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sodium Bicarbonate (NaHCO3) (Active Comparator): In this double-blind, crossover-designed study, 19 recreational female runners will be randomly assigned to either a bicarbonate or a placebo group.
  Interventions: Dietary Supplement: Sodium Bicarbonate (NaHCO3)
- Sodium Chloride (Placebo Comparator): Each participant will complete two trials: acute SB and placebo. A dose of 0.3 g/kg/day SB will be administered in 7 ml/kg water with a carbohydrate-rich meal to minimize gastrointestinal (GIS) symptoms.
  Interventions: Dietary Supplement: Sodium Chloride

INTERVENTIONS:
Dietary Supplement: Sodium Bicarbonate (NaHCO3) — Participants will complete two interventions: sodium bicarbonate (SB) and placebo (PL). In the SB condition, participants will receive 0.3 g/kg SB, while in the PL condition, they will receive 0.03 g/kg table salt, administered double-blind.
  Arms: Sodium Bicarbonate (NaHCO3)
Dietary Supplement: Sodium Chloride — Participants will complete two interventions: sodium bicarbonate (SB) and placebo (PL). In the SB condition, participants will receive 0.3 g/kg SB, while in the PL condition, they will receive 0.03 g/kg table salt, administered double-blind.
  Arms: Sodium Chloride

SUMMARY:
Sodium bicarbonate (SB) is one of the ergogenic aids that enhance short-duration, high-intensity sports performance by improving the buffering system. However, studies suggest that SB may also be beneficial for prolonged high-intensity endurance exercises, where anaerobic glycolysis plays a role. The commonly used SB dose in these studies (0.3 g/kg) often leads to gastrointestinal (GI) discomfort, necessitating alternative approaches. Among various protocols, consuming SB with a carbohydrate-rich meal has been identified as an effective strategy to mitigate GI distress. Although some studies indicate a positive effect of SB on performance, research involving female athletes remains limited, comprising only 7.4% of the total studies. Given that women generally have lower muscle mass and fewer type II muscle fibers, their glycolytic capacity might be lower, and SB could have distinct physiological effects on them. While SB has been shown to enhance anaerobic performance in female athletes, its impact on high-intensity endurance exercise performance has not yet been investigated. This study aims to examine the effects of acute sodium bicarbonate ingestion, consumed with a carbohydrate-rich meal, on prolonged high-intensity running performance, acid-base balance, and GI response in female runners. In this double-blind, crossover-designed study, 19 recreational female runners will be randomly assigned to either a bicarbonate or a placebo group. The bicarbonate group will ingest 0.3 g/kg SB, while the placebo group will consume 0.03 g/kg salt, both 90 minutes before exercise, alongside a carbohydrate-rich meal. Participants will then complete a 10 km time-trial run, aiming for their best performance. Throughout the study, GI symptoms, exercise completion time, blood lactate, pH, bicarbonate levels, heart rate, and perceived exertion during exercise will be assessed. Performance tests will be conducted twice during the follicular phase of the menstrual cycle, with a 3-7 days washout period between trials. A two-way repeated measures ANOVA will be used to compare the effects of the interventions.

DETAILED DESCRIPTION:
Introduction Buffering Agents in Exercise Performance During high-intensity exercise, muscle fatigue occurs, negatively impacting both anaerobic and aerobic (endurance) exercise performance. One primary cause of muscle fatigue is metabolic acidosis, which arises from the accumulation of intracellular lactate and H+ ions (Freis et al., 2017; Krustrup et al., 2015). Since muscle acidity is regulated by intracellular and extracellular buffering systems, enhancing these systems is essential to sustain effective muscle contraction, delay fatigue, and thereby optimize performance in both anaerobic and high-intensity endurance exercises (Durkalec-Michalski et al., 2018a; 2018b).

Various ergogenic aids are utilized to boost intracellular and extracellular buffering capacity, with beta-alanine and sodium bicarbonate (SB) being two well-supported agents: Beta-alanine enhances intracellular buffering by increasing muscle carnosine levels, thereby preventing acidosis and improving performance (Trexler et al., 2015). SB primarily acts as an extracellular buffer, clearing H+ ions from the blood. This mechanism indirectly reduces H+ accumulation in muscles during intense exercise (Durkalec-Michalski et al., 2018a; 2018b). By preserving ATP production via glycolysis, this buffering action delays the onset of muscle fatigue during high-intensity exercises (Lancha Junior et al., 2015; Lopes-Silva et al., 2019).

Due to its ability to reduce lactate and H+ accumulation, research has predominantly focused on SB's effects on high-intensity, short-duration exercise (1-10 minutes) performance reliant on glycolytic metabolism (Delextrat et al., 2018; Driller et al., 2012; Gough et al., 2017). For example, 0.3 g/kg dose of SB intake improved total work output by enhancing buffering capacity in a 10 x 6-second sprint protocol (Miller et al., 2016). SB is thus commonly used for sports reliant on glycolytic metabolism, such as sprinting, middle-distance running, and combat sports. Additionally, SB may also be beneficial for longer endurance events (30-60 minutes) at the anaerobic threshold (AT), such as high-intensity interval training or long-distance endurance events concluding with a final sprint (Burke, 2013).

SB and Endurance Performance While long-duration endurance exercise (>30 minutes) is primarily driven by aerobic metabolism, anaerobic glycolysis also significantly contributes to energy production, leading to elevated blood lactate levels (Egger et al., 2014; Jones et al., 1977; McNaughton et al., 1999). Consequently, SB can help maintain optimal pH levels during endurance exercise, enhancing high-intensity performance at or near the aerobic threshold (Egger et al., 2014; Freis et al., 2017).

Studies have examined the effects of 0.2-0.3 g/kg SB intake on endurance performance near the lactate threshold in cycling and running, often comparing it to neutral (sodium chloride) or acidic (ammonium chloride) supplements. Findings indicate that while SB improves time to exhaustion, acidic agents can reduce it (George & MacLaren, 1988; Jones et al., 1977; Sutton et al., 1981). For instance, Egger et al. (2014) found that 0.3 g/kg SB intake one hour before exercise extended performance time during a test following a 30-minute exercise session at 95% anaerobic threshold.

While studies have supported SB's positive effects on endurance performance, there is mixed evidence. Some studies found that, despite increasing blood bicarbonate and pH or reducing lactate levels, SB did not improve endurance performance (Freis et al., 2017; McNaughton et al., 1999). These studies, however, were conducted under laboratory conditions. Research on SB's effect in field-based, real-world endurance settings has not yet been conducted.

Optimizing Sodium Bicarbonate Intake While SB has shown promise in enhancing high-intensity endurance performance, studies often focus on acute SB usage, typically recommending a 0.3 g/kg dose before exercise (Lancha Junior et al., 2015). This protocol effectively increases blood pH and bicarbonate levels (Price & Singh, 2008) while reducing plasma H+ concentration (Renfree, 2007). However, this acute intake can lead to gastrointestinal symptoms (GIS) due to the rapid absorption of both bicarbonate and sodium (Siegler et al., 2012). In endurance sports, managing GIS is critical, as such symptoms can more severely impact performance than in short-duration events (Jeukendrup, 2017).

This has prompted the exploration of alternative SB protocols to minimize GIS, such as spreading the dosage over time, using lower doses, or administering over consecutive days. In a study conducted by researchers involved in this project, the effects of 0.2 g/kg SB on endurance performance were evaluated over four consecutive days in male cyclists. The results showed that while both acute and consecutive SB intake enhanced buffering capacity (Figure 1), only consecutive intake significantly extended time to exhaustion compared to placebo (Figure 2). Notably, GIS was observed with acute intake but was minimized with consecutive-day intake, suggesting the need for alternative acute SB protocols to further improve endurance performance by reducing GIS.

Figure 1. Effects of 0.2 g/kg Sodium Bicarbonate on Blood pH (A) and Blood Bicarbonate Levels (B) on Acute and Consecutive Days (Aktitiz et al., 2024). SB: Sodium Bicarbonate. §: Significant difference between Acute SB and PLA (p < 0.05); ¥: Significant difference among all pairwise comparisons (Acute SB, Consecutive Days SB, and PLA) (p < 0.05).

Figure 2. Effect of 0.2 g/kg Sodium Bicarbonate on Time to Exhaustion on Acute and Consecutive Days (Aktitiz et al., 2024). SB: Sodium Bicarbonate. *: Significant difference between Consecutive Days SB and PLA (p < 0.05).

In studies on alternative SB intake methods, consumption with carbohydrate-rich meals was found to be one of the most effective ways to prevent GIS. For instance, a study (Carr et al., 2011) showed that consuming 0.3 g/kg SB with 1.5 g/kg carbohydrate and 7 ml/kg fluid resulted in peak blood bicarbonate and pH levels within 120-150 minutes, with minimal GIS. This finding suggests that SB consumption with carbohydrates may enhance performance while minimizing adverse effects, providing a promising approach for endurance athletes.

SB and Female Athletes Although studies have demonstrated that SB can positively impact high-intensity endurance exercise performance (Egger et al., 2014; George & MacLaren, 1988; Jones et al., 1977; Sutton et al., 1981), most research has been conducted on male athletes. Studies involving female athletes represent only 7.4% of the total SB studies (Smith et al., 2022). Due to their generally lower muscle mass and a reduced proportion of type 2 muscle fibers (Nuzzo et al., 2024), women may have reduced glycolytic capacity, meaning SB could have a distinct effect on female physiology (Green et al., 1984; Hegge et al., 2016; Janssen et al., 2000; Porter et al., 2002). Additionally, due to their monthly experience with gastrointestinal symptoms (GIS) such as bloating, abdominal pain, and diarrhea during the menstrual cycle, women may tolerate SB's side effects better (Carr et al., 2023). These findings suggest that SB might be more effective in female athletes.

Indeed, an acute dose of 0.3 g/kg SB taken 90 minutes before exercise was shown to enhance 1-minute maximal cycling performance in 10 physically active women (McNaughton et al., 1997). In another study involving female basketball players (n=15), a 3-day regimen of 0.4 g/kg SB improved repeated sprint performance and jump height during a simulated game (Delextrat et al., 2018). A meta-analysis also confirmed SB's positive effect on anaerobic performance in female athletes (Saunders et al., 2022). However, the impact of SB on high-intensity endurance performance in female athletes has not been investigated. Furthermore, existing studies are limited to highly trained women aged 19-26 (Saunders et al., 2022), and its effects on recreational-level and older female athletes remain unexplored.

In summary, while significant evidence suggests that SB can enhance high-intensity endurance performance, there is a notable lack of research specifically addressing female athlete physiology and alternative SB protocols that mitigate GIS in women.

METHOD Study Group The study will include 19 healthy female recreational runners aged 18-40, who have been consistently training (at least three days per week) for a minimum of one year. Participants will be recruited through outreach to university sports clubs in Ankara. Ethics approval for this study was obtained from the Hacettepe University Clinical Research Ethics Committee. Participants will be informed of the protocol, provided with informed consent forms, and the study will adhere to the updated Declaration of Helsinki (2013). Demographic forms documenting training history and an American College of Sports Medicine Physical Activity Readiness Questionnaire will be administered to confirm eligibility.

Inclusion Criteria:

* Female, aged 18-40.
* Recreational runner with a minimum one-year history of regular training (at least three days per week).
* Experience in races of 10 km or more (verified by an official race result).
* Ability to complete a 10 km distance at an average pace below 6.00 min/km (confirmed through best-record evidence via applications like Strava).

Exclusion Criteria:

* Usage of any medications or supplements that could impact metabolism.
* Presence of any acute or chronic condition limiting physical activity (musculoskeletal, cardiovascular, or respiratory issues).
* Alcohol and/or smoking habits.
* Adherence to a specific diet influencing metabolism during the study period (intermittent fasting, ketogenic, vegan diets, etc.).
* Pregnancy or breastfeeding during the study period.
* Severe menstrual irregularities or amenorrhea.
* Body Mass Index (BMI) outside the range of 18.5-30.
* History of gastrointestinal disorders (e.g., IBS, Crohn's disease).
* Allergy or intolerance to sodium bicarbonate or related compounds.
* History of disordered eating.

Study Design This randomized, double-blind, crossover study will involve each participant in four experimental exercise tests: one for body composition, one maximal oxygen uptake (VO2max) test, and two "performance tests" focused on evaluating 10 km completion time and other endurance-related variables. Participants will complete two interventions: sodium bicarbonate (SB) and placebo (PL). In the SB condition, participants will receive 0.3 g/kg SB, while in the PL condition, they will receive 0.03 g/kg table salt, administered double-blind. Performance testing will commence 1.5 hours after ingestion of a standardized 1.5 g/kg carbohydrate breakfast. After each test, a washout period of 3-7 days will occur, after which the groups will be crossed over, and the protocol repeated.

Body Composition Participants will visit the laboratory after an overnight fast, wearing no metal or electronic items, and will void their bladders before measurements. Body weight will be measured to a precision of 0.1 kg using an electronic scale (Tanita UBB SC 330, USA). Body composition, including fat mass, body fat percentage, lean body mass, and visceral adipose tissue, will be assessed using Dual-energy X-ray Absorptiometry (DXA, Lunar Prodigy Pro narrow Fan Beam, GE Health Care, Madison Wisconsin, USA). The DXA will be calibrated daily, and all measurements will be conducted by a licensed researcher. Body composition values will be analyzed using GE Encore v14.1 software and CoreScan for visceral adipose tissue.

Standardization of Dietary Intake One day of dietary intake records will be collected 24 hours before performance tests and analyzed using the BEBIS 6.1 software (Stuttgart, Germany). This standardization will ensure similar carbohydrate intake before tests. Additionally, participants will consume a standardized 1.5 g/kg carbohydrate breakfast (cereal, milk, fruit) 90 minutes before testing, aligning with race-day recommendations (Burke et al., 2011).

Sodium Bicarbonate Supplementation Each participant will complete two trials: acute SB and placebo. A dose of 0.3 g/kg/day SB will be administered in 7 ml/kg water with a carbohydrate-rich meal to minimize gastrointestinal (GIS) symptoms, following the protocol by Carr et al. (2011). For placebo, 0.03 g/kg/day table salt will be administered at the same intervals. Participants' GIS symptoms will be evaluated using a 10-point Likert scale survey assessing 10 different GIS symptoms at 90, 60, and 30 minutes pre-exercise.

VO2max

To determine participants' VO2max and fitness levels, an incremental treadmill test protocol will be conducted. The test will begin at 6 km/h and increase by 1 km/h each minute until exhaustion, with a treadmill incline set to 1%. Oxygen uptake (VO2) and carbon dioxide production (VCO2) will be measured using a gas analysis system (Quark CPET, Cosmed Cardio-Pulmonary Exercise Testing, Italy), and heart rate will be monitored using a Polar Ignite and H9 sensor. The VO2max value will be considered valid if two of the following criteria are met:

* A plateau in VO2.
* Respiratory exchange ratio >1.10.
* Heart rate exceeding 90% of the predicted max.
* Perceived exertion score above 18. 10 km Run Performance Test To assess the impact of SB on prolonged high-intensity exercise, participants will perform a 10 km time trial following a warm-up routine of 5 minutes jogging at 8 km/h and 5 minutes stretching. Participants will be instructed to avoid exercise 2 days before, abstain from alcohol (48 hours) and caffeine (12 hours), and maintain their usual diet. Tests will be conducted at the same time, under similar environmental conditions, in the follicular phase (days 6-12) of the menstrual cycle to minimize hormonal impact (McNulty et al., 2020). Participants will be asked to report their menstrual cycle phase and oral contraceptive use during test scheduling.

Participants will be informed that they are expected to deliver their best performance. During their first visit, participants will be asked to verify their previous fastest 10 km performance using an application. For each performance trial, the percentage relative to their previous personal best 10 km performance will be calculated to assess their actual performance. Participants will be asked to consume 5-10 ml/kg of water 2-3 hours before the test, and the amount of fluid intake will be recorded to ensure the same amount is consumed during the second visit. Urine samples will be collected before the performance test to evaluate urine specific gravity using a refractometer (Atago Digital Urine S.G. UG-α alpha), with values assessed as follows: ≤1.020 for euhydration, 1.020-1.030 for hypohydration, and >1.030 for severe hypohydration. To calculate the percentage of fluid loss, body weight will be measured before and after exercise. The difference between pre- and post-exercise body weight will be adjusted for the amount of fluid consumed during the exercise, and the percentage of fluid loss will be calculated by dividing this value by the initial body weight. Proper hydration will be ensured by evaluating water intake, urine specific gravity, and fluid loss percentage to control hydration's effect on performance.

No additional foods, aside from the standardized meal, will be consumed on the morning of the test. Water intake during the test will be unrestricted, but the amount consumed will be recorded to ensure similar intake in subsequent tests. During the test, blood samples will be taken from the fingertip before the test begins and at the 1st, 3rd, 5th, and 7th minutes after the test ends to measure blood pH, lactate, and bicarbonate levels. Heart rate (HR) will be continuously monitored using a heart rate monitor (Polar Ignite Heart Rate Monitor and Polar H9 Heart Rate Sensor, Polar Electro Inc., USA), and real-time HR data will be tracked by the researcher. Participants will be verbally informed of the completion of each kilometer, but no feedback will be provided regarding HR, speed, or time, and no verbal encouragement will be given. Performance data will be shared with participants only after all measurements are completed.

To avoid bias, all measurements for the same participant will be conducted by the same researcher, and the researcher administering the performance test will be blinded to the sodium bicarbonate (SB) or placebo randomization. The performance time obtained at the end of the test will serve as the primary performance outcome for the study. In addition to the 10 km completion time and speed, the time and speed for every 400 m, the first 1 km, 1-5 km, 5-9 km, last 1 km, and final 400 m will also be evaluated. The perceived exertion at the end of the test will be assessed using the BORG scale (6-20 points).

Blood Sampling and Analysis Blood samples will be collected from the fingertip at baseline and at 1, 3, 5, and 7 minutes post-exercise to analyze blood pH, bicarbonate, lactate, pO2, and pCO2 using a blood gas analyzer (ABL 9, Radiometer, Germany).

Data Analysis Sample size calculations performed using G*Power software (version 3.1.9.2) indicate a minimum of 19 participants is required for a power of 90% at an alpha level of 0.05 with an effect size of 0.8. Data will be analyzed with SPSS 23.0, presented as means ± standard deviations, and tested for normality using the Shapiro-Wilk test. Repeated Measures ANOVA will analyze performance times, while a Two-Way Repeated Measures ANOVA will assess blood parameters (intervention x time). Significance is set at p<0.05. Bonferroni post hoc tests will identify significant differences, and partial eta squared (ƞ²) will be calculated to determine effect sizes (ƞ² ≤ 0.01 = small, ƞ² ≤ 0.06 = medium, ƞ² ≤ 0.14 = large) (Richardson, 2011).

ELIGIBILITY:
Inclusion Criteria:

* Female, aged 18-40.
* Recreational runner with a minimum one-year history of regular training (at least three days per week).
* Experience in races of 10 km or more (verified by an official race result).
* Ability to complete a 10 km distance at an average pace below 6.00 min/km (confirmed through best-record evidence via applications like Strava).

Exclusion Criteria:

* Usage of any medications or supplements that could impact metabolism.
* Presence of any acute or chronic condition limiting physical activity (musculoskeletal, cardiovascular, or respiratory issues).
* Alcohol and/or smoking habits.
* Adherence to a specific diet influencing metabolism during the study period (intermittent fasting, ketogenic, vegan diets, etc.).
* Pregnancy or breastfeeding during the study period.
* Severe menstrual irregularities or amenorrhea.
* Body Mass Index (BMI) outside the range of 18.5-30.
* History of gastrointestinal disorders (e.g., IBS, Crohn's disease).
* Allergy or intolerance to sodium bicarbonate or related compounds.
* History of disordered eating.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Estimated)
Dates: Start 2024-11-03 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
10 km time-trial run | 1 year
  To assess the impact of SB on prolonged high-intensity exercise, participants will perform a 10 km time trial following a warm-up routine of 5 minutes jogging at 8 km/h and 5 minutes stretching.Participants will be informed that they are expected to deliver their best performance. During their first visit, participants will be asked to verify their previous fastest 10 km performance using an application. For each performance trial, the percentage relative to their previous personal best 10 km performance will be calculated to assess their actual performance. The performance time obtained at the end of the test will serve as the primary performance outcome for the study. In addition to the 10 km completion time and speed, the time and speed for every 400 m, the first 1 km, 1-5 km, 5-9 km, last 1 km, and final 400 m will also be evaluated.

SECONDARY OUTCOMES:
blood gas parameters | 1 year
  Blood samples will be collected from the fingertip at baseline and at 1, 3, 5, and 7 minutes post-exercise to analyze blood pH, bicarbonate, lactate, pO2, and pCO2 using a blood gas analyzer.

OTHER OUTCOMES:
gastrointestinal (GIS) symptoms | 1 year
  Participants' GIS symptoms will be evaluated using a 10-point Likert scale survey assessing 10 different GIS symptoms at 90, 60, and 30 minutes pre-exercise.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
At this stage, no final decision has been made regarding the sharing of individual participant data (IPD). We will update our IPD sharing plan.

REFERENCES:
- [Background] Carr AJ, McKay AKA, Burke LM, Smith ES, Urwin CS, Convit L, Jardine WT, Kelly MK, Saunders B. Use of Buffers in Specific Contexts: Highly Trained Female Athletes, Extreme Environments and Combined Buffering Agents-A Narrative Review. Sports Med. 2023 Dec;53(Suppl 1):25-48. doi: 10.1007/s40279-023-01872-7. Epub 2023 Oct 25. PMID 37878211
- [Background] Aktitiz S, Kosar SN, Turnagol HH. Effects of acute and multi-day low-dose sodium bicarbonate intake on high-intensity endurance exercise performance in male recreational cyclists. Eur J Appl Physiol. 2024 Jul;124(7):2111-2122. doi: 10.1007/s00421-024-05434-1. Epub 2024 Feb 29. PMID 38421429